CLINICAL TRIAL: NCT01478295
Title: Effectiveness of Nursing Intervention on Quality of Life of Older Caregivers: Clinical Trial Randomised by Clusters
Brief Title: Effectiveness of Nursing Intervention on Caregivers
Acronym: CuidaCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Milagros Rico Blazquez, Nurse, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FIS PI11/02132
Record Dates: First submitted 2011-11-15; First posted 2011-11-23 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Quality of Life
Keywords: Nursing intervention; Primary Health care; caregiver; strain
MeSH Terms: conditions — Sprains and Strains | interventions — Methods; Primary Health Care; Caregivers; Quality of Life; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CuidaCare Intervention (Experimental): Regular care in consultation or home and Structured nursing care (CuidaCare intervention): improved strategies for coping, health education on self-care and dependent care and emotional support. 10 visits are structured, with a periodicity of approximately 2 visits per month and last for 30 to 40 minutes each
  Interventions: Behavioral: CuidaCare Intervention; Other: Control Group/Usual Care:
- Control Group/Usual Care (Active Comparator): Usual care in consultation or home, which is to respond to the specific demands of care of the caregiver, using the resources of the nursing discipline.
  Interventions: Other: Control Group/Usual Care:

INTERVENTIONS:
Behavioral: CuidaCare Intervention — Nursing intervention address to Caregiver Standardized care plan (PCE) Coping strategies promoting social support and empowerment through health education
  Other Names: Nursing intervention; Primary Health care; Caregiver; Strain; Quality of life; Standardized care plan (PCE)
  Arms: CuidaCare Intervention
Other: Control Group/Usual Care: — Control Group/Usual Care:
  Standardized care plan (PCE) Coping strategies promoting social support and empowerment through health education

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a structured nursing intervention (PCE), including two types of intervention defined in the literature (coping strategies promoting social support and empowerment through health education), which has an effect on the perceived quality of life for the caregiver, when compared with conventional intervention or non-support.

DETAILED DESCRIPTION:
Aim: to compare the effectiveness of a standardized care plan (SCP) compared to the usual nursing intervention to improve the quality of life for primary caregivers over 65 years old measured through points change with the EuroQol-5D (EQ-5D) scale.

Secondary objectives:

Evaluate the influence of prognostic variables on quality of life of caregiver. Describe the level of caregiver burden. Describe the socio-demographic profile of the dependent person and caregiver.

Method:

Design: cluster randomized trial. Setting: study in Health Centers Primary Care of Area of Madrid Health Service. Subjects: unit of randomization: primary healthcare centres. Analysis unit: caregivers over 65 years old.

Intervention: The SCP in the treatment group and the usual intervention in the control group.

Sample size adjusted for design effect= 218 (109 in each arm). Main response variable: perceived quality of life (EQ-5D). Secondary response variables: nursing diagnosis, Zarit Caregiver Burden Interview, objective overload level.

Prognostic variables:Dependent person-related: dependence level (Barthel, Lawton-Brody), cognitive dysfunction (Pfeiffer).

Caregiver-related: depression scale (Yesavage), anxiety level (Goldberg), family function (family Apgar). Sociodemographic variables.

Data Analysis: Analysis of main effectiveness by intention to treat, comparing the difference in units on the EQ-5D scale before and post- intervention in both groups at 0, 6, 12 and 18 months. The estimation adjusted, using logistic regression with aleatory effects, those data that can act as confounding factors or change the effect.

ELIGIBILITY:
Inclusion Criteria:

* Not psychological treatment or social support during the study period.
* Be able to follow the trial's demands.
* Experience of caring for at least 6 months in a year.
* Caregivers who consent to take part.

Exclusion Criteria:

* Caregivers of patients hospitalized during the initial data collection.
* Caregivers of institutionalized patients.
* Severe psychiatric conditions including depression and major affective pictures.
* Paid caregivers.
* Experience as a caregiver for less than a month.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 266 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Perceived quality of life | Change from baseline in quality of life at 18 months after the intervention
  Perceived quality of life: Quality of life measured by EuroQol (EQ5D) Scale Change from baseline in quality of life at 18 months after the intervention

SECONDARY OUTCOMES:
Nursing diagnosis | Change from Baseline in Nursing diagnosis at 18 months after the intervention
  Use NANDA International Classification to measure: caregiver role strain or caregiver role (risk for) or stress(overload).
  Change from Baseline in Nursing diagnosis at 18 months after the intervention
Caregiver Burden | Change from Baseline in Caregiver Burden at 18 months after the intervention
  Zarit Caregiver Burden Interview. Change from Baseline in Nursing diagnosis at 18 months after the intervention.
Depression scale | Change from Baseline in Depression scale at 18 months after the intervention
  Yesavage Depression scale. Change from Baseline in Depression scale at 18 months of the intervention.
Anxiety level | Change from Baseline in Anxiety level at 18 months after the intervention
  Goldberg scale. Change from Baseline in Anxiety level at 18 months after the intervention
Family function | Change from Baseline in Family function at 18 months after the intervention
  Family Apgar test. Change from Baseline in Family function at 18 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Rico, Nurse, Principal Investigator — Gerencia Atención Primaria. Madrid
Locations (1):
- Gerencia Atención Primaria, Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Background] Rico-Blazquez M, Escortell-Mayor E, Del-Cura-Gonzalez I, Sanz-Cuesta T, Gallego-Berciano P, de Las Casas-Camara G, Soto-Diaz S, Garcia-Sanz P, Harris-de-la-Vega N, Martin-Martin M, Dominguez-Perez L, Rivera-Alvarez A, Sarrion-Bravo JA, Perez-de-Hita C, de-Frias-Redondo M, Ferrer-Arnedo C, Hernandez-Pascual M, Valdivia-Perez A, Farina YR. CuidaCare: effectiveness of a nursing intervention on the quality of life's caregiver: cluster-randomized clinical trial. BMC Nurs. 2014 Jan 27;13(1):2. doi: 10.1186/1472-6955-13-2. PMID 24467767
- [Derived] Rico-Blazquez M, Quesada-Cubo V, Polentinos-Castro E, Sanchez-Ruano R, Rayo-Gomez MA, Del Cura-Gonzalez I; CuidaCare Group. Health-related quality of life in caregivers of community-dwelling individuals with disabilities or chronic conditions. A gender-differentiated analysis in a cross-sectional study. BMC Nurs. 2022 Mar 29;21(1):69. doi: 10.1186/s12912-022-00845-x. PMID 35351100